CLINICAL TRIAL: NCT00855231
Title: Diagnostic Accuracy of Multislice CT Angiography for Acute Chest Pain - Assessment of Chest Pain Utilizing a Triple Rule Out Evaluation With Computed Tomography (ACUTE CT) Trial
Brief Title: Diagnostic Accuracy of Multislice CT Angiography for Acute Chest Pain
Acronym: ACUTE CT
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Kelley Branch, Assistant Professor, University of Washington
Other Study IDs: 27903-D; 05-6337-D 03
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Chest Pain; Acute Coronary Syndrome; Pulmonary Embolism; Aortic Dissection
Keywords: Acute coronary syndrome; Coronary artery disease; cardiac imaging; computed tomography
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome; Pulmonary Embolism; Aortic Dissection; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The ACUTE CT trial is designed to test whether the assessment of chest structures by high-resolution multislice computed tomography (CT) provides equivalent diagnostic accuracy for patient with acute chest pain or other potential cardiac symptoms as compared to a standard of care evaluation.

DETAILED DESCRIPTION:
Adults at low to intermediate risk of acute coronary syndrome who present to the Emergency Department with symptoms suggestive of cardiac ischemia will undergo a blinded cardiac CT followed by a standard of care (SOC) strategy. Significant coronary artery disease on CT (coronary stenosis >50%) will be compared to an adjudicated diagnosis derived from clinical data and other diagnostic tests based on the SOC strategy. Costs for the SOC evaluation will be collected and compared to a CT-based evaluation. Patients will be followed for 3 years after enrollment to evaluate prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Low to intermediate risk of angina with a TIMI ACS Risk Score ≤ 4
* chest pain or other symptoms suggestive of ACS within 24 hours
* male ≥30 years or female ≥45 years old
* at least one cardiac risk factor
* no obvious cause for symptoms.

Exclusion Criteria:

* known CAD
* ST segment elevation, new left bundle branch block or dynamic ECG changes
* creatinine ≥1.8 g/dL
* pregnant or lactating female
* hemodynamic or respiratory instability
* ongoing bronchospasm
* known iodinated contrast allergy
* atrial fibrillation or irregular heart rate

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Alll patients presenting to the University of Washington Medical Center Emergency Department with possible acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2006-07; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of CT compared to standard of care evaluation | 3 months

SECONDARY OUTCOMES:
Cost savings of CT-based evaluation compared to the standard of care evaluation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kelley R Branch, MD, Principal Investigator — University of Washington; William P Shuman, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Branch KR, Busey J, Mitsumori LM, Strote J, Caldwell JH, Busch JH, Shuman WP. Diagnostic performance of resting CT myocardial perfusion in patients with possible acute coronary syndrome. AJR Am J Roentgenol. 2013 May;200(5):W450-7. doi: 10.2214/AJR.12.8934. PMID 23617513
- [Background] Branch KR, Strote J, Shuman WP, Mitsumori LM, Busey JM, Rue T, Caldwell JH. Diagnostic accuracy and clinical outcomes of ECG-gated, whole chest CT in the emergency department. PLoS One. 2013 Apr 16;8(4):e61121. doi: 10.1371/journal.pone.0061121. Print 2013. PMID 23613797
- [Background] Branch KR, Bresnahan BW, Veenstra DL, Shuman WP, Weintraub WS, Busey JM, Elliott DJ, Mitsumori LM, Strote J, Jobe K, Dubinsky T, Caldwell JH. Economic outcome of cardiac CT-based evaluation and standard of care for suspected acute coronary syndrome in the emergency department: a decision analytic model. Acad Radiol. 2012 Mar;19(3):265-73. doi: 10.1016/j.acra.2011.10.029. Epub 2011 Dec 30. PMID 22209422
- [Result] May JM, Shuman WP, Strote JN, Branch KR, Mitsumori LM, Lockhart DW, Caldwell JH. Low-risk patients with chest pain in the emergency department: negative 64-MDCT coronary angiography may reduce length of stay and hospital charges. AJR Am J Roentgenol. 2009 Jul;193(1):150-4. doi: 10.2214/AJR.08.2021. PMID 19542407
- [Result] Shuman WP, Branch KR, May JM, Mitsumori LM, Strote JN, Warren BH, Dubinsky TJ, Lockhart DW, Caldwell JH. Whole-chest 64-MDCT of emergency department patients with nonspecific chest pain: Radiation dose and coronary artery image quality with prospective ECG triggering versus retrospective ECG gating. AJR Am J Roentgenol. 2009 Jun;192(6):1662-7. doi: 10.2214/AJR.08.1872. PMID 19457832
- [Result] Mitsumori LM, Wang E, May JM, Lockhart DW, Branch KR, Dubinsky TJ, Shuman WP. Triphasic contrast bolus for whole-chest ECG-gated 64-MDCT of patients with nonspecific chest pain: evaluation of arterial enhancement and streak artifact. AJR Am J Roentgenol. 2010 Mar;194(3):W263-71. doi: 10.2214/AJR.09.2788. PMID 20173125
- [Result] Shuman WP, May JM, Branch KR, Mitsumori LM, Strote JN, Green DE, Caldwell JH. Negative ECG-gated cardiac CT in patients with low-to-moderate risk chest pain in the emergency department: 1-year follow-up. AJR Am J Roentgenol. 2010 Oct;195(4):923-7. doi: 10.2214/AJR.09.3972. PMID 20858819